CLINICAL TRIAL: NCT04408989
Title: A Randomized, Double-Blind, Three-Arm, Single Dose, Parallel Study To Compare the Pharmacokinetics, Safety and Immunogenicity of MB02-SP, MB02-DM (Bevacizumab Biosimilar Drugs) and US-licensed Avastin® in Healthy Male Volunteers
Brief Title: A Study Comparing the Pharmacokinetic Similarity of MB02-SP, MB02-DM and US Licensed-Avastin®.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MB02-A-06-20
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MB02-SP (Bevacizumab Biosimilar) (Experimental): Sterile vial 100mg/4ml, single-dose 1mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: MB02-SP
- MB02-DM (Bevacizumab Biosimilar) (Experimental): Sterile vial 100mg/4ml, single-dose 1mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: MB02-DM
- US licenced Avastin® (Active Comparator): Sterile vial 100mg/4ml, single-dose 1mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: US licenced Avastin®

INTERVENTIONS:
Drug: MB02-SP — Solution for intravenous infusion, single dose of 1mg/kg, administered as 90-minute infusion
  Other Names: MB02-SP (Bevacizumab Biosimilar)
  Arms: MB02-SP (Bevacizumab Biosimilar)
Drug: MB02-DM — Solution for intravenous infusion, single dose of 1mg/kg, administered as 90-minute infusion
  Other Names: MB02-DM (Bevacizumab Biosimilar)
  Arms: MB02-DM (Bevacizumab Biosimilar)
Drug: US licenced Avastin® — Solution for intravenous infusion, single dose of 1mg/kg, administered as 90-minute infusion
  Other Names: Bevacizumab (US sourced)
  Arms: US licenced Avastin®

SUMMARY:
Randomized, double blind, parallel group, single dose, 3 arm study to investigate and compare the PK, safety and immunogenicity profile of MB02-DM with MB02-SP and US-Avastin® in healthy male subjects.

During the course of the study, the similarity in pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms. Safety, tolerability, and immunologic response to the administered drugs will also be evaluated throughout.

DETAILED DESCRIPTION:
The primary PK parameter endpoints are Cmax and AUC0-∞ for bevacizumab. The secondary PK endpoints will include all other PK parameters for bevacizumab, including tmax, t1/2, CL and AUC(0-t).

The serum PK parameters of bevacizumab will be calculated using standard noncompartmental methods. An analysis of covariance model will be used to analyse the log-transformed primary PK parameters (AUC[0 ∞] and Cmax) and AUC(0-t). The model will include a fixed effect for treatment and body weight as a covariate.

All other PK parameters will not be subject to inferential statistical analysis.

Estimates of geometric mean ratios together with the corresponding 90% confidence intervals (CI) will be derived for the comparisons of the PK parameters as follows:

* MB02-SP versus MB02-DM
* MB02-SP versus US Avastin®
* MB02-DM versus US Avastin®

PK similarity will be achieved if the 90% CIs for the biosimilar-to-reference ratios of PK endpoints (AUC[0-∞] and Cmax) fall within the predefined 0.80-1.25 acceptance similarity criteria for all 3 pairwise comparisons; MB02-SP versus MB02-DM; MB02-SP versus US Avastin®; and MB02-DM versus US Avastin®.

All AEs will be listed and summarised using descriptive methodology. All observed or patient-reported AEs will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The incidence of AEs for each treatment will be presented by severity and by association with the study drugs as determined by the Investigator (or designee). Each AE will be coded using the Medical Dictionary for Regulatory Activities. All safety data will be listed and summarised as appropriate.

Immunogenicity data (overall ADA incidence and titters, and neutralising ADA results) will be listed. A summary of the number and percent of subjects testing positive for ADA or neutralising antibodies before the dose of MB02-SP, MB02-DM, or US Avastin® (Day -1) and at scheduled post dose assessments will be presented by treatment arm. All safety data and immunogenicity data summaries will be based on the safety analysis population. Select analyses may be repeated for subsets with or without ADA and de novo ADA formation as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Males of any race, between 18 and 55 years of age, inclusive, at Screening.
2. Body mass index between 18.5 and 29.9 kg/m2, inclusive, at Screening.
3. Total body weight between 50 and 95 kg, inclusive, at Screening.
4. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital non-haemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is acceptable) at Screening or Check-in as assessed by the Investigator (or designee).
5. Relevant clinical laboratory evaluations of haematology, coagulation, urinalysis and clinical chemistry within normal range at Screening and Check in as follows. A single repeat test will be allowed at each timepoint.

   * Absolute neutrophil count ≥1.5 × 109 L
   * Platelet count ≥100 × 109 L
   * Haemoglobin >10 g/dl
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 x ULN
   * Alkaline phosphatase (ALP) ≤1.5 × ULN
   * Total bilirubin <1.5 × ULN (<51.30 µmol/L in subjects with Gilbert's syndrome)
   * Blood urea nitrogen ≤1.5 × ULN
   * Creatinine <132.63 µmol/L
   * Serum albumin: >35 g/L
   * Low density lipoprotein cholesterol ≤ 4.9 mmol/L
   * High density lipoprotein cholesterol ≥ 0.85 mmol/L
   * Creatine kinase (CK) <2 × ULN
   * International normalised ratio (INR) 0.8 to 1.3
   * Urine dipstick for proteinuria <2+
6. Systolic blood pressure ≥90 mmHg and <140 mmHg and diastolic blood pressure ≥50 mmHg and <90 mmHg at Screening and Check in.
7. Subjects agree to use contraception.
8. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions. Subjects must have signed an informed consent before any study-related procedure or evaluation is performed.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. Any current or recent history of active infections, including localised infections (Within 2 months prior Screening Visit for any serious infection which requires hospitalization or intravenous anti-infective, and within 14 days prior Screening Visit for any active infection which requires oral treatment).
4. History of, or planned surgery, including suturing, dental surgery or wound dehiscence within 30 days of dosing, or within 30 days of the last study visit.
5. Presence of a nonhealing wound or fracture.
6. Known history of clinically significant essential hypertension, orthostatic hypotension, fainting spells or blackouts for any reason, cardiac failure or history of thromboembolic conditions.
7. Medically significant dental disease or dental neglect, with signs and/or symptoms of local or systemic infection that would likely require a dental procedure during the course of the study.
8. Clinically relevant history of alcoholism, addiction or drug/chemical abuse prior to Check-in, and/or positive alcohol breath test and/or urinary drug test screen (confirmed by repeat) at Screening or Check in.
9. History of bleeding disorders or protein C, protein S, and/or factor V Leiden deficiency.
10. History of clinically significant haemorrhage, epistaxis, GI bleeding, haemorrhoids and/or haemoptysis.
11. History of GI perforation, ulcers, gastro oesophageal reflux, inflammatory bowel disease, diverticular disease, or any fistulae.
12. Alcohol consumption of >24 units per week. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
13. Positive hepatitis panel, positive human immunodeficiency test. Subjects whose results are compatible with prior immunisation and not infection may be included at the discretion of the Investigator.
14. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to Check-in, or within 5 half lives of the investigational drug used in the study.
15. Use or intend to use slow-release medications/products considered to still be active within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
16. Use or intend use of any prescription medications/ nonprescription products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator or designee.
17. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
18. Have received a live or attenuated vaccine from 3 months prior to Screening or have the intention to receive a vaccine during the study.
19. Intend to travel to a region where a vaccination will be required due to endemic disease within 3 months of dosing.
20. Previous treatment with an anti VEGF antibody or any other protein or antibody targeting the VEGF receptor.
21. Use of tobacco- or nicotine-containing products within 1 year prior to Check-in, or positive cotinine test upon Screening or Check-in.
22. Receipt of blood products within 60 days prior to Check-in.
23. Donation of blood from 90 days prior to Screening, plasma from 14 days prior to Screening, or platelets from 42 days prior to Screening.
24. Poor peripheral venous access.
25. History of abnormal peripheral sensation including paraesthesia and/or numbness in arms and/or legs.
26. Have previously completed or withdrawn from this study or any other study investigating bevacizumab, and/or have previously received bevacizumab.
27. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.
28. Vulnerable subjects (e.g. persons kept in detention).
29. Subjects who are study site employees or immediate family members of a study site or Mabxience employee.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects may be enrolled
Enrollment: 114 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schwabe, MD, Principal Investigator — Auckland Clinical Studies; Alexandra Cole, MD, Principal Investigator — Christchurch Clinical Studies
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Christchurch Clinical Studies Trust, Christchurch

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Started | 37 | 39 | 38
Completed | 37 | 39 | 35
Not Completed | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin® | Total
Number analyzed (Participants) | 37 | 39 | 38 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (11.15) | 30.8 (10.44) | 34.1 (10.68) | 32.04 (10.76)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Only male subjects | 37 | 39 | 38 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 0 | 0 | 2 | 2
  White | 23 | 27 | 27 | 77
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 5 | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.94 (2.396) | 24.34 (2.162) | 24.79 (2.786) | 24.68 (2.47)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) - (AUC[0-∞])
Description: Compare the pharmacokinetic (PK) profiles of the 3 arms (AUC[0-∞])
Time Frame: Pre-dose (0 hours),end of infusion, 2, 3, 4, 5, 6, 7, 12, and 24 hours and at Days 3, 4, 5, 6, 7, 8, 10, 14, 21, 28, 42, 56, 78, and 100 post-dose
Population: The PK population included all subjects who received the full dose of MB02-SP, MB02-DM or US-Avastin®, did not had any major protocol deviations, and had evaluable PK data for at least one timepoint
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Number analyzed (Participants) | 37 | 39 | 38
h*ng/ml | 7500000 (12.3) | 8000000 (15.8) | 7520000 (14.4)
Statistical Analysis 1: Comparison: MB02-SP (Bevacizumab Biosimilar) vs MB02-DM (Bevacizumab Biosimilar); Test type: Equivalence — PK similarity was achieved if the 90% CIs for the biosimilar-to-reference ratios of AUC(0-∞) were within the predefined 0.80-1.25 acceptance similarity criteria. The PK parameter AUC(0-∞) was log-transformed (base e) prior to analysis and was analysed using an ANCOVA model. The model included treatment as a fixed effect and body weight as a covariate; Ratio of GLSM = 0.943, 90% CI 2-sided [0.899 to 0.989] — For the comparison, MB02 SP represents the numerator and MB02 DM represents the denominator
Statistical Analysis 2: Comparison: MB02-SP (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of GLSM = 1.00, 90% CI 2-sided [0.956 to 1.05] — For the comparison, MB02 SP represents the numerator and US Avastin represents the denominator
Statistical Analysis 3: Comparison: MB02-DM (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of GLSM = 1.07, 90% CI 2-sided [1.01 to 1.12] — For the comparison, MB02 DM represents the numerator and US Avastin represents the denominator

2. Primary Outcome: Pharmacokinetics (PK) - (Cmax)
Description: Compare the pharmacokinetic (PK) profiles of the 3 arms (Cmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Number analyzed (Participants) | 37 | 39 | 38
ng/ml | 25600 (15.7) | 27400 (14.9) | 26100 (16.6)
Statistical Analysis 1: Comparison: MB02-SP (Bevacizumab Biosimilar) vs MB02-DM (Bevacizumab Biosimilar); Test type: Equivalence — PK similarity was achieved if the 90% CIs for the biosimilar-to-reference ratios of Cmax were within the predefined 0.80-1.25 acceptance similarity criteria. The PK parameter Cmax was log-transformed (base e) prior to analysis and was analysed using an ANCOVA model. The model included treatment as a fixed effect and body weight as a covariate; Ratio of GLSM = 0.937, 90% CI 2-sided [0.887 to 0.989] — For the comparison, MB02 SP represents the numerator and MB02 DM represents the denominator
Statistical Analysis 2: Comparison: MB02-SP (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 0.983, 90% CI 2-sided [0.925 to 1.05] — For the comparison, MB02 SP represents the numerator and US Avastin represents the denominator
Statistical Analysis 3: Comparison: MB02-DM (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.05, 90% CI 2-sided [0.991 to 1.11] — For the comparison, MB02 DM represents the numerator and US Avastin represents the denominator

3. Secondary Outcome: Other PK Parameters (Tmax)
Description: Evaluation of all other PK parameters (tmax) tmax = time of maximum observed serum concentration
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Number analyzed (Participants) | 37 | 39 | 38
hours | 4.02 [1.50 to 8.00] | 5.00 [1.50 to 6.30] | 5.00 [1.52 to 12.00]

4. Secondary Outcome: Other PK Parameters (AUC[0 t])
Description: Evaluation of all other PK parameters (AUC[0 t]) AUC(0-t) = AUC from time zero to the time of last quantifiable concentration
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Number analyzed (Participants) | 37 | 39 | 38
h*ng/ml | 7010000 (14.8) | 7550000 (16.9) | 7110000 (15.4)

5. Secondary Outcome: Other PK Parameters (CL)
Description: Evaluation of all other PK parameters (CL) CL = total body clearance of drug after intravenous administration
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Number analyzed (Participants) | 37 | 39 | 38
L/h | 0.0103 (13.9) | 0.00975 (15.2) | 0.0104 (16.5)

6. Secondary Outcome: Other PK Parameters (t1/2)
Description: Evaluation of all other PK parameters (t1/2) t½ = apparent serum terminal elimination half-life
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Number analyzed (Participants) | 37 | 39 | 38
hours | 390 (17.2) | 393 (11.1) | 396 (14.4)

7. Secondary Outcome: Immunogenicity
Description: Number of participants with anti-bevacizumab antiboides (ADA), including neutralizing antibodies (Nab).
  Subjects who tested positive at baseline are not included here.
Time Frame: Days -1, 14, 28, 56 and 78
Population: The safety population included all subjects exposed to MB02-SP, MB02-DM or US-Avastin®, and had at least one post dose safety assessment
Measure: Number; unit: participants
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Number analyzed (Participants) | 37 | 39 | 38
participants
  ADA positive | 8 | 13 | 9
  nAb positive | 0 | 0 | 0

8. Secondary Outcome: Safety (Number of Participants Reporting Treatment-related Adverse Events)
Description: Number of participants who reported Treatment-related Adverse Events using the CTCAE v5.0 criteria
Time Frame: Day 1 - Day 100
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Number analyzed (Participants) | 37 | 39 | 38
Participants
  Subjects with TEAEs | 24 | 23 | 29
  Subjects with SAEs | 0 | 0 | 0
  Subjects discontinued due to TEAEs | 0 | 0 | 0
  Deaths | 0 | 0 | 0

9. Secondary Outcome: Safety (Treatment-related Adverse Events)
Description: Treatment-related Adverse Events based on the CTCAE v5.0 criteria reported by the study participants
Time Frame: Day 1 - Day 100
Population: as for outcome 7
Measure: Number; unit: events
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
Number analyzed (Participants) | 37 | 39 | 38
events
  TEAEs | 42 | 58 | 59
  Related TEAEs (possibly, probably and related TEAES) | 12 | 9 | 6
  Unrelated TEAES (unlikely and not related) | 30 | 49 | 53
  Mild (Grade 1) TEAES | 39 | 55 | 50
  Moderate (Grade 2) TEAES | 3 | 3 | 9
  Severe (Grade 3) TEAES | 0 | 0 | 0
  Life-Threatening (Grade 4) TEAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study duration (Day 1 - Day 100)
Description: Coded according to Medical Dictionary for Regulatory Activities (version 24.0), and graded on the basis of the US National Cancer Institute's Common Terminology for Adverse Events (version 5.0).
Arm/Group | MB02-SP (Bevacizumab Biosimilar) | MB02-DM (Bevacizumab Biosimilar) | US Licenced Avastin®
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 14/37 | 22/39 | 24/38
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MB02-SP (Bevacizumab Biosimilar) (N=37) | MB02-DM (Bevacizumab Biosimilar) (N=39) | US Licenced Avastin® (N=38)
Headache (Nervous system disorders) | 3 (3) | 6 (7) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 3 (4)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Catheter site bruise (General disorders) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT04408989/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT04408989/SAP_001.pdf